CLINICAL TRIAL: NCT00551408
Title: The Determination of Endothelial Progenitor Cells in Pulmonary Idiopathic Arterial Hypertension.
Brief Title: Endothelial Progenitor Cells and Pulmonary Idiopathic Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Unidad de Investigacion Clinica en Medicina S.C. (Network)
Responsible Party: Principal Investigator, Dr. Carlos jerjes-Sanchez Diaz, Principal investigator, Unidad de Investigacion Clinica en Medicina S.C.
Other Study IDs: UDICEM07-012; 07-012
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Idiopathic Arterial Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: 20 patients with idiopathic pulmonary arterial hypertension in the WHO functional class II to III, and had a mean pulmonary artery pressure >30 mm Hg on right heart catheterization able to walk >50 m during a standardized 6-min walk test.

SUMMARY:
Endothelial dysfunction ultimately represents an imbalance between the magnitude of injury and the capacity for repair.

Current evidence established that endothelial progenitor cells (EPC) participate in several models of vascular disease as acute coronary syndromes, stroke, diabetes, peripheral artery disease, etc. However EPC in the setting of PAH is less well established. The target of this study is to demonstrate if the number of EPC is increased in a mexican population of patients with PAH.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included in the study if they were in The WHO functional class II to III, and had a mean pulmonary artery pressure >30 mm Hg on right heart catheterization. The ability to walk >50 m during a standardized 6-min walk test.

Exclusion Criteria:

* Pulmonary hypertension as a result of heart disease, pulmonary disease, sleep-associated disorders, chronic thromboembolic disease, autoimmune or collagen vascular disease, HIV infection, liver disease, major bleeding requiring blood transfusion,renal dysfunction, and evidence for malignant diseases were excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IPAH between 18 and 70 years of age of either gender were invited to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos J Sanchez Diaz, MD., Principal Investigator — Unidad de Investigacion Clinica en Medicina SC.
Locations (1):
- Unidad de Investigacion Clinica en Medicina SC., Monterrey, Nuevo León, Mexico